CLINICAL TRIAL: NCT02172391
Title: The Effects of Tiotropium Therapy on Airway Diameter in Patients With COPD (a Randomized, Double-blind, Placebo-controlled, Parallel-group Study)
Brief Title: Effect of Tiotropium on Airway Diameter in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.218
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Tiotropium (Experimental): Tiotropium inhalation powder capsules 18 mcg, one capsule once daily for 28 days
  Interventions: Drug: Tiotropium inhalation powder capsules
- Placebo (Placebo Comparator): Placebo inhalation powder capsules, one capsule once daily for 28 days
  Interventions: Drug: Placebo inhalation powder capsules

INTERVENTIONS:
Drug: Tiotropium inhalation powder capsules
  Arms: Tiotropium
Drug: Placebo inhalation powder capsules
  Arms: Placebo

SUMMARY:
Trial to investigate the acute and chronic effect of tiotropium therapy on airway diameter in COPD patients as measured by inspiratory capacity (IC).

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of chronic obstructive pulmonary disease
* Male or female patients ≥ 40 years of age but ≤ 75 years old
* Patients must have a smoking history of more than ten pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes per day for a year
* Patients must be able to perform all specified procedures and maintain records during the study period as required in the protocol
* Patients must be able to inhale medication from the HandiHaler®
* All patients must sign a Patient Informed Consent Form prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications
* Patients must be willing to attend an outpatient clinic on a regular basis
* Patients must be able to walk 164 feet (50 meters) during the Six Minute Walk Test

Exclusion Criteria:

* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis test results, if the abnormality defines a disease listed as an exclusion criterion
* Patients with a serum glutamic-oxaloacetic transaminase (SGOT) ≥1.5 x Upper Limit of Normal Range (ULN), serum glutamic-pyruvic transaminase (SGPT) ≥1.5 x ULN, bilirubin ≥1.5 x ULN or creatinine ≥ 1.5 x ULN regardless of the clinical condition
* Patients with a recent history (i.e., one year or less) of myocardial infarction
* Patients with a recent history (i.e., three years or less) of heart failure, pulmonary edema or patients with any cardiac arrhythmia (with or without symptoms)
* Patients with regular use of daytime oxygen therapy
* Patients with known active tuberculosis
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history or a thoracotomy for other reason should be evaluated as per exclusion criterion no. 1
* Patients with upper respiratory tract infection in the past six weeks prior to the Screening Visit or during the baseline period
* Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients who are being treated with cromolyn sodium or nedocromil sodium
* Patients who are being treated with antihistamines (H1 receptor antagonists) or antileukotrienes and are not able to stop these medications 1 month before visit 1
* Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception
* Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥ 600/mm3
* Patients with history of (past five years or less) and/or active alcohol or drug abuse
* Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Period (Visit 1)
* Patients who have participated in any pulmonary rehabilitation program for COPD within 6 weeks prior to Visit 1 or throughout the study
* Limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea such as arthritis in the leg, angina or claudication

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81
Dates: Start 2000-11; Primary Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 to 3 hours (AUC0-3) of resting inspiratory capacity (IC) | Day 28
Trough resting IC | Day 28

SECONDARY OUTCOMES:
FEV1 (Forced expiratory volume in one second) | Day 1, 14 and 28
FVC (forced vital capacity) | Day 1, 14 and 28
FEF25%-75% (Forced Expiratory Flow, mid expiratory phase) | Day 1, 14 and 28
FEF50% (Forced Expiratory Flow, at 50% of FVC) | Day 1, 14 and 28
FEF75% (Forced Expiratory Flow, at 75% of FVC) | Day 1, 14, 28
SVC (Slow vital capacity) | Day 1, 14, 28
Respiratory System Transfer Impedance (Respiratory Resistance) | Day 1, 14 and 28
Airway Resistance (Raw) | Day 1, 14 and 28
Thoracic Gas Volume (TGV) | Day 1, 14 and 28
Specific Airway Conductance (SGaw) | Day 1, 14 and 28
Physician's Global Evaluation | Day 1 and 28
Oxygen Saturation (SaO2) prior to six minute walk test | Day 1 and 28
Oxygen Saturation (SaO2) post six minute walk test | Day 1 and 28
IC prior to six minute walk test | Day 1 and 28
IC post six minute walk test | Day 1 and 28
Chronic Respiratory Questionnaire (CRQ) | Day 1 and 28
Baseline Dyspnea Index (BDI) | Day 1
Transition Dyspnea Index (TDI) | Day 28
Change from baseline in seated blood pressure | Baseline, Day 1, 14 and 28
Change from baseline in pulse rate | Baseline, Day 1, 14 and 28
Occurrence of Adverse Events | until day 35